CLINICAL TRIAL: NCT05199051
Title: AGORA-1 /ALFA 2100 Study : A Phase 2 Study of Gemtuzumab Ozogamicin (GO)-Gilteritinib Combination in Adults With FLT3-ITD and/or FLT3-TKD Relapse/Refractory (R/R) AML
Brief Title: A Phase 2 Study of Gemtuzumab Ozogamicin (GO)-Gilteritinib Combination in Adults With FLT3-ITD and/or FLT3-TKD Relapse/Refractory (R/R) AML
Acronym: AGORA-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Collaborators: Astellas Pharma Inc (Industry); Pfizer (Industry); Acute Leukemia French Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/65; 2023-504176-25-00 (EU CTIS Number); 2021-001813-35 (EudraCT Number)
Record Dates: First submitted 2021-11-12; First posted 2022-01-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: AML; Leukaemia (Acute Myeloid)
Keywords: AML; Gemtuzumab Ozogamicin Gilteritinib Combination; relapse; refractory; Leukaemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemtuzumab ozogamicine - Cytarabine - Gilteritinib (Experimental): For Gemtuzumab ozogamicine administrated during the induction phase at D1, D4 and D7, 3mg/m2/day (5mg max), IV, 2h of infusion.
  For Cytarabine during induction and consolidation phase at D1 to D5, 1000 mg/m2, IV, 2h of infusion.
  For Gilteritinib during induction phase from D10 for 14 consecutive days, per os, two doses level study with dose level 1 (80mg/d) in part 1 or dose level 2 (80 or 120mg/d depending of the result of part 1) in part 2.
  During consolidation (2 cycles max) from D8 for 14 consecutive days, per os, 120mg/d or reduced dose of 80 mg/kg is planned to be used in patients receiving concomitantly CYP3A4 inhibitors.
  During the maintenance (24 months max) dose level 2 (120mg/d), per os.
  Interventions: Combination Product: Gemtuzumab ozogamicine - Cytarabine - Gilteritinib

INTERVENTIONS:
Combination Product: Gemtuzumab ozogamicine - Cytarabine - Gilteritinib — See Arms description paragraph
  Other Names: Mylotarg - Aracytine - Xospata

SUMMARY:
This is a national, open-label, single-arm, multicenter phase II trial evaluating the safety and efficacy of adding gilteritinib, a new FLT3 inhibitor to the AGORA platform, consisting of the combination of an intermediate dose of cytarabine and a divided dose of GO in adult patients with R / R AML with an FLT3-ITD and/or FLT3-TKD mutation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or more
* Confirmed diagnosis of R/R AML positive for CD33 antigen as determined locally by immunophenotyping according to routine practice, defined as:

  * AML refractory to 1 or 2 intensive chemotherapy courses or a treatment by hypomethylating agents (HMAs)
  * Or AML in first hematologic relapse or progression after front-line therapy, including intensive chemotherapy or hypomethylating agents (HMAs).
  * Previous treatments with FLT3 inhibitors (other than gilteritinib) are allowed
  * R/R AML secondary to a prior chemotherapy or radiotherapy for another cancer (tAML) could be included.
* Presence of a FLT3-ITD mutation (allelic ratio ≥0.05 at last evaluation)* or a FLT3 TKD mutation
* Patient with no contraindication to gemtuzumab ozogamicin (GO), cytarabine and gilteritinib
* ECOG performance status ≤2
* AST and ALT ≤ 2.5 x upper the limit of normal (ULN) and/or total and direct serum bilirubin ≤ 1.5 x ULN unless considered due to leukemia
* Estimated glomerular filtration rate (GFR) ≥ 50 mL/min according to the formula usually used by the investigator
* Written informed consent obtained prior to any screening procedures
* Eligible for National Health Insurance in France

Exclusion Criteria:

* Acute promyelocytic leukemia or AML with BCR-ABL1 gene fusion
* Secondary AML (sAML) defined by a history of prior myelodysplastic syndrome (MDS) or myeloproliferative syndrome (MPN) including chronic myelomonocytic leukemia (CMML)
* Patient with contraindications to the administration of gemtuzumab ozogamicin (GO), cytarabine and gilteritinib. Refer to the SPCs of the molecules mentioned concerning the contraindications, special warnings, precautions for use, dose modifications in the event of toxicity, contraception and monitoring of patients and drugs prohibited or to be used with caution.
* Proven central nervous system leukemic involvement
* Prior allogeneic HSCT within the last 6 months and/or history of acute GVHD of grade >1
* Prior treatment with gemtuzumab ozogamicin within the last 3 months preceding the initiation of the treatment in the present clinical trial
* Uncontrolled or active malignant disease within prior 12 months (excluding cutaneous basal cell carcinoma, "in-situ" carcinoma of the cervix or breast, or other local malignancy excised)
* Uncontrolled or significant cardiovascular history or symptoms including:

  * Prior anthracycline exposure equivalent to more than 550 mg/m2 of daunorubicin
  * History of clinically relevant ventricular arrhythmias (e.g. ventricular tachycardia, ventricular fibrillation or torsade de pointes)
  * History of 2° (Mobitz II) or 3° heart block (subjects with pacemakers are allowed if they have no history of clinically relevant arrhythmias with the pacemaker)
  * History of uncontrolled angina pectoris or MI within 6 months
  * History of NYHA Class 3 or 4 heart failure
  * Left ventricular ejection fraction ≤ 50% or less than the institutional lower limit of normal
  * History of complete left bundle branch block
  * Unstable angina, New York Heart Association (NYHA) class 3 or 4 congestive heart failure
  * QTcF > or equal to 450 msec, long QT syndrome (including family history)
  * Bradycardia < 50 bpm (unless subject has a pacemaker)
  * Systolic BP ≥ 180 mmHg or diastolic BP ≥ 110 mmHg
* Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate treatment)
* Active known HBV or HCV hepatitis or positive HIV serology
* Concurrent therapy with any other investigational agent or cytotoxic drug, within 28 days before starting treatment. Only hydroxyurea ± dexamethasone is permitted for the control of blood counts
* Current use or anticipated requirement for drugs that are known strong inducers of CYP3 A4/5
* Current use or anticipated requirement for drugs that are known as strong inhibitors or inducers of P glycoprotein (P-gp), as mentioned in the appendix 14 of the protocol, with the exception of drugs that are considered absolutely essential for the care of the subject
* Current use or anticipated treatment with concomitant drugs that target 5HT1R or 5HT2BR receptors or sigma non-specific receptor, as mentioned in the appendix 15 of the protocol, with exception of drugs that are considered absolutely essential for the care of the subject
* Known malabsorption syndrome or other condition that may significantly impair absorption of oral study medications
* Any of concurrent severe and/or uncontrolled medical condition, which could compromise participation in the study.
* Patient currently receiving one or more inadvisable or prohibited treatments described in section 6.4.2 of the protocol.
* Females who are pregnant or breastfeeding.
* Women of childbearing potential or partners of women of childbearing potential should use a highly effective method of contraception during treatment and change the duration of contraception after the last dose of the medicines of the study (GO, cytarabine and gilteritinib).

  * For women of childbearing potential (WOCBP): agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception with a failure rate of < 1% per year during the treatment period and after the final dose of study treatment for at least: - 7 months for GO, - 6 months for cytarabine, - 6 months for gilteritinib. Women must refrain from donating eggs during this same period. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization is permanently infertile due to surgery (i.e. removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Hormonal contraceptive methods must be supplemented by a barrier method. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. If required per local guidelines or regulations, locally recognized acceptable methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form. Women of childbearing potential must have a negative serum pregnancy test result within 7 days prior to first dose.
  * For male patients: acceptance that most of the study treatments require specific reliable and effective contraception measures, as well as measures related to sperm donation Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating sperm, as defined below With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and after the final dose of study treatment for at least: - 4 months for GO, - 6 months for cytarabine, - 4 months for gilteritinib.

Men must refrain from donating sperm during this same period With pregnant female partners, men must remain abstinent or use a condom to avoid exposing the embryo during the treatment period and for at least: - 4 months for GO, - 6 months for cytarabine, - 4 months for gilteritinib. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. If required per local guidelines or regulations, locally recognized acceptable methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

* Adults subject to a legal protection order or unable to give their consent
* Persons deprived of their freedom by judicial or administrative decision, persons hospitalized without their consent by virtue of articles L. 3212-1 and L. 3213-1 and who are not subject to the provisions of article L. 1121-8.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2028-07-10 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Stage 1 - Safety of the addition of gilteritinib to the AGORA treatment platform | 18 months
  The primary objective of the first stage is to evaluate the safety of combining gilteritinib with the Gemtuzumab Ozogamicin (GO) -cytarabine AGORA platform in patients with FLT3-ITD and/or FLT3-TKD mutated Relapse/Refractory (R/R) Acute Myeloïd Leukemia (AML), through occurrence of dose-limiting toxicity (DLT).
Stage 2 - Event-free survival (EFS) | 60 months
  The primary objective of the second extension stage is to evaluate the efficacy of combining gilteritinib with the Gemtuzumab Ozogamicin (GO)-cytarabine AGORA platform in patients with FLT3-ITD and/or FLT3-TKD mutated Relapse/Refractory (R/R) Acute Myeloïd Leukemia (AML) through event-free survival (EFS).

SECONDARY OUTCOMES:
Response rates to the study treatment | 60 months
  Response rate, including Complete Response (CR), Incomplete Hematologis Recovery (CRi) and partial hematologic recovery (CRh)*; the overall response rate (ORR) being defined as CR/CRi/CRh rates
  *: CRi, CR with incomplete hematologic recovery, meaning CR with platelet count <100,000/µL or absolute neutrophil count <1000/µL; CRh, CR with partial hematologic recovery, meaning CR not fulfilling CR or CRi criteria but with platelet count >50,000/µL AND absolute neutrophil count >500/µL.
Early mortality rates, at day-30 | 30 months
  Mortality rates between day 1 and day 30
Incidence of subsequent allogeneic Hematopoietic Stem Cell Transplantation (HSCT) overall. | 60 months
  Incidence of subsequent allogeneic HSCT of all patients of the study.
Incidence of subsequent allogeneic Hematopoietic Stem Cell Transplantation in responding patients specifically. | 60 months
  Incidence of subsequent allogeneic HSCT in responding patients specifically.
Evaluation of Duration of response (DOR) of treatment | 60 months
  Duration of response (DOR).
Evaluation of relapse-free survival (RFS) | 60 months
  Duration of relapse-free survival (RFS) of patient.
Evaluation of overall survival (OS) | 60 months
  Duration of overall survival (OS) defined as the time between the date of the inclusion and the date of death or the date of last news for those still alive at the end of the follow-up.
Subgroup analyses defined by patient | 60 months
  Subgroups defined by a patient related factor: age (<65 vs ≥65y)
Subgroup analyses defined by disease | 60 months
  Subgroups defined by disease related factors: cytogenetics, mutation profiles (including NPM1 and FLT3-ITD), ELN-risk classification 2017.
Subgroup analyses defined by allograft | 60 months
  Subgroups defined by treatment related factor by the performance of a subsequent allogeneic HSCT.
Evaluation of the Safety : incidence of SAE (SAEs) | 60 months
  Safety through Serious Adverse event (SAEs)
Evaluation of the Safety : incidence of Adverses Events (AEs) | 60 months
  Safety through Adverse event (AEs), Serious Adverse event (SAEs), Treatment Emergent Adverse Event (TEAEs) and incidence of sinusoidal obstruction syndrome (SOS))
Evaluation of the Safety : incidence of Treatment Emergent Adverse Event (TEAEs) | 60 months
  Safety through Treatment Emergent Adverse Event (TEAEs)
Evaluation of the Safety : incidence of sinusoidal obstruction syndrome (SOS) | 60 months
  Safety through incidence of sinusoidal obstruction syndrome (SOS)

CONTACTS AND LOCATIONS:
Overall Officials: Juliette LAMBERT, MD-PHD, Principal Investigator — Versailles Hospital
Locations (12):
- France (12):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - CHMS de Chambery, Chambéry
  - HIA Percy, Clamart
  - CHU Limoges, Limoges
  - CHRU Nancy, Nancy
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hôpital Saint Louis, Paris
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier de Versailles, Versailles